CLINICAL TRIAL: NCT06992349
Title: Evaluating the Efficacy of Bioptron° Light Therapy in Managing Primary Dysmenorrhea Among Obese Adolescence: Double Blinded Randomized Control Trial
Brief Title: Bioptron Light Therapy for Dysmenorrhea in Obese Adolesences: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Noureldeen Kora (Other)
Responsible Party: Sponsor-Investigator, Alaa Noureldeen Kora, Principal Investigator, Sinai University
Organization: Sinai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU.REC.2024 (26 H)
Record Dates: First submitted 2025-02-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Dysmenorrhea Primary; Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: women with BMI more than 30 and receive active bioptron© (Experimental)
  Interventions: Device: bioptron light therapy
- Group 2: women with BMI between 18.5 to 25 and receive active bioptron©. (Experimental)
  Interventions: Device: bioptron light therapy

INTERVENTIONS:
Device: bioptron light therapy — BIOPTRON® Hyperlight is a proprietary, optimized blend of visible and infrared light properties that Bio-stimulate cells and speeding up the healing process of a wide range of medical diseases.
  Bioptron© light therapy has been utilized as a non-invasive treatment for wound healing, skin ulcers, and various musculoskeletal conditions(Abd Elhamid et al., 2020).

SUMMARY:
Dysmenorrhea is the most common health problem in women in the reproductive age(Bakhsh et al., 2022). The primary dysmenorrhea starts shortly after the menarche the pain lasting 1 to 3 days that start just before or at the onset of menstruation with the absence of other gynecological symptoms (Itani et al., 2022). Primary dysmenorrhea can reduce the quality of life and social activities of women(Esan et al., 2024).

There is a relationship between body mass composition and primary dysmenorrhea and as the value of body mass index and body fat percentages goes on increasing in females, the severity of primary dysmenorrhea also increased (Wu et al., 2022).

BIOPTRON® Light therapy system is a device that contains an optical unit. This unit emits light with an electromagnetic spectrum produced by the sun, but without the ultraviolet rays and it is significant with four main characteristics which are Polarization, Polychromatic, Incoherence and low energy light (Raeissadat et al., 2014).

The Purpose of the Study The aim of the study is to investigate the effect of bioptron© light therapy on primary dysmenorrhoea outcomes as pain and quality of life among obese adolescence.

ELIGIBILITY:
Inclusion Criteria:

* 144 female adolescences suffering from primary dysmenorrhea pain determined according to the sample size calculation adapted from (Gu et al., 2022).
* They will be selected from the outpatient's clinic of the faculty of Physical Therapy Sinai University.
* Their chronological age ranged from 16 to 18 years old.

Exclusion Criteria:

* Those who were taking anti-psychotic or anti-depressant medications, patients with any skin lesion or infection.
* Gynecological disorders included cervical cancer, ovarian tumors, endometriosis, uterine fibroids, polycystic ovarian syndrome, and other conditions that can affect menstruation.

Ages: 16 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
number of anatomical pain locations, pain range, number of days of pain during menstruation (and frequency of disabling pain to perform their activities. | At the end of Cycle 1 (each cycle is 28 days)".

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS): is a single-item question that asks the patient to rate the pain on a scale of 0 to 10. | At the end of Cycle 1 (each cycle is 28 days)".
Algometer is an objective measurement of the degree of pressure required to evoke a painful response over selected trigger points. | At the end of Cycle 1 (each cycle is 28 days)".
The EuroQol-5 Dimension (EQ-5D), developed in 1990, is a most widely used generic tool to measure health-related quality of life. | At the end of Cycle 1 (each cycle is 28 days)".

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No